CLINICAL TRIAL: NCT06780072
Title: The Acute Effect of Manual Massage Therapy on Daytime Napping in Poor Sleepers
Brief Title: Impact of Massage on Daytime Napping
Acronym: TakeAnap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Nicosia (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2094-2/08-02-2023
Record Dates: First submitted 2025-01-10; First posted 2025-01-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Sleep Deprivation
Keywords: Massage; day-time nap; poor sleepers; PSG; Relaxation; power naps
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned into 3 conditions each one week apart: 1) the control condition (CON) where subjects will not receive any intervention, while they were rested for 35 min on a massage bed; 2) the activation condition (ACT) where subjects will receive an activation (Sports) massage session lasting for 30 min and rested for 5 min without any interference; and 3) the relaxation condition (REL) where subjects will receive a relaxation massage session lasting for 30 min and rested for 5 min without any interference (Figure 2). All conditions will be separated by one week apart and take place at the exact time of the day, while the order of the various conditions will be randomly assigned.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): For the control condition (CON) participants will not receive any intervention, while they will be rested for 35 min on a massage bed
- Activation Massage (Experimental): For the activation condition (ACT) participants will receive an activation (Sports) massage session lasting for 30 min and rest for 5 min without any interference.
  Interventions: Other: Activation Massage therapy
- Relaxation Massage (Experimental): For the relaxation condition (REL) participants will receive a relaxation massage session lasting for 30 min and rest for 5 min without any interference.
  Interventions: Other: Relaxation Massage Therapy

INTERVENTIONS:
Other: Activation Massage therapy — Massage Sessions
  Activation (Sports) massage The activation (sports) type of massage will be used as one of the massage interventions. This technique will be performed on a full body with more attention given to specific leg muscle groups such as the feet, the gastrocnemius, the femoral biceps and quadriceps and in upper body muscle groups such as the triceps, the rhomboid, the deltoid, the trapezius and head areas. Briefly, this type of massage involves a wide range of techniques that include effleurage, palmar sliding, pounding and hacking. The total duration of the activation message will be 30 minutes.
  Arms: Activation Massage
Other: Relaxation Massage Therapy — Relaxation massage The Relaxation type of massage will be used as the second type of intervention in this study. This technique is designed to promote deep relaxation, reduce stress and enhance overall well-being. It is characterized by the use of four primary techniques performed on the full body, including the palms and feet. Specifically, these techniques consist of effleurage
  Arms: Relaxation Massage

SUMMARY:
In the quest for optimal physical and mental performance and recovery, people are constantly exploring various strategies to enhance their overall well-being. Daytime napping helps mitigate the effects of inadequate nighttime sleep, allowing people to reduce fatigue and potentially improve physical performance. Research has also shown that strategically timed naps can significantly boost athletic performance, improve cognitive function, and reduce daytime fatigue.

Short naps lasting between 10 to 60 minutes are ideal for quickly boosting alertness and cognitive function. Additionally, they can facilitate a complete sleep cycle, including REM sleep, which is crucial for both physical and mental recovery. Massage therapy, recognized for its ability to alleviate muscle soreness, improve circulation, and induce relaxation and it might play a crucial role in facilitating a good night sleep.

In athletes a massage therapy serves as both a proactive and reactive measure in optimizing sports and exercise performance, ensuring athletes are physically and mentally prepared for competition while also facilitating their recovery, minimizing the risk of injury and being particularly effective in alleviating pain. Massage therapy significantly contributes to improving night sleep efficiency as well as the duration of sleep onset.[12] From a biochemical point of view, massage promotes the release of serotonin, a hormone that enhances the sense of wellbeing. In addition, serotonin is a biosynthetic precursor of melatonin and an active neurotransmitter, whose levels affect various functions of the body including sleep promotion,[14] while can play a significant role in mental health as it regulates mood and emotional well-being.

Nowadays, massage has evolved into various types that are specialized for the treatment of various health problems. The most well know and frequently used types of massage are the "sports massage" and the "relaxation massage". Sports massage has been proven to enhance athletic performance, as well as help athletes recover after competition while the Deep Relaxation massage is used exclusively for the relaxation and psychological discharge. More specifically, the relaxation-therapeutic massage uses pressure that is deeply relaxing, but not painful, smooth gliding strokes that are both rhythmic and flowing, which increases blood circulation and promotes a general sense of relaxation. Even thought, these 2 very common types of massage have been applied for many years in various settings, it is not clear whether massage affects brain function and state of alertness.

Therefore, the primary aim of the current study is to investigate the effect of two different types of manual massage sessions on daytime napping using objective (EEG - brain activity) and subjective (questionnaires) measurements of relaxation in poor sleepers.

DETAILED DESCRIPTION:
The current study will assess the impact of two different massage styles in aspects related to relaxation and wakefulness using a polysomnography system and questionnaire measurements.

The volunteers of the current study will participate in 3 different scenarios, each 5 days apart: Scenario 1 is the control session when participants will lay down on the prone position on a professional massage bed for 35 min without any interventions, Scenario 2 will be the experimental session 1 where participants will lay down on the prone position on a professional massage bed for 35 min receiving a deep relaxation massage session, and Scenario 3 will be the experimental session 2, where participants will lay down on the prone position on a professional massage bed for 35 min receiving a Activation/Stimulation type of massage session. During all three scenarios participants' brain signal and subjective perceived feeling of relaxation will be recorded. Scenario 2 and 3 are taking place in a random order in every participant.

Materials and Methods Subjects Fifteen (N=15) participants will be included in the current study. Inclusion criteria include subjects of both sexes, aged >18 years, and Pittsburgh Quality Sleep Index score >5. Exclusion criteria include a history of mental illness, dermatological diseases, allergies to massage oil, history of epilepsy and any acute or chronic condition that would limit the ability of the patient to participate in the study.

Study Design Subjects will randomly be assigned into 3 conditions each one week apart: 1) the control condition (CON) where subjects will not receive any intervention, while they are rested for 35 min on a massage bed; 2) the activation condition (ACT) where subjects will receive an activation (Sports) massage session lasting for 30 min and rest for 5 min without any interference; and 3) the relaxation condition (REL) where subjects receive a relaxation massage session lasting for 30 min and rest for 5 min without any interference (Figure 2). All conditions will be separated one week apart and take place at the exact time of the day, while the order of the various conditions is randomly assigned. All massage sessions were delivered by a professional masseur, while the researchers analyzing the data will be blind to the assigned group. All measurements will be conducted at the sleep laboratory under controlled conditions, with a constant room temperature of 22°C. The study is approved by the Human Research and Ethics Committee of the University of Thessaly (2094-2/08-02-2023). All Subjects will give their written informed consent prior to study participation.

Procedure All measurements will be performed in the Lifestyle Medicine Laboratory, at the Department of Physical Education and Sports Science of Trikala, in Thessaly, Greece.

Before the initiation of the study, subjects will complete a series of questionnaires and measurements related to overall health. Subjects will be connected to a portable polysomnographic EEG/EOG system (HST-mit-tablet, SOMNOmedics AG, Randersacker, Germany) for the recording of brain activity. Before and after each condition, subjects will complete a relaxation sensation questionnaire (RSQ) for assessing the state of relaxation and perform 3 maximum handgrip attempts to assess the level of muscle strength. Measurements of vital signs such as resting heart rate and blood pressure also will be recorded. The participants will be free to either sleep or stay awake during the whole intervention period.

Measuring Instruments Body Composition Body composition will be assessed using anthropometric measurements including BMI, and bioimpedance (Tanita DC-360 S, Serinth) under standard methodology.

Questionnaires The following questionnaires will be administered using the interview method by experienced researchers.

* The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality and the existence of any sleep abnormalities.
* The Short Form survey 36-item 36 quality of life questionnaire (SF-36) will be used to assess the quality of life.
* The Beck Depression Inventory (BDI) questionnaire will be used to assess depressive symptoms and signs.
* The Perceived Stress Scale (PSS) will be used to assess the level of stress.
* The Relaxation State Questionnaire (RSQ) will be used to assess the state of relaxation.

Brain Activity / Arousal Assessment The Home Sleep Test (HST) (www.somnomedics.de), will be used to assess brain activity during napping periods. This is a portable sleep monitoring system that enables the recording of various sleep parameters in a natural setting, as the patient's bedroom. EEG signals will be analyzed in 30 sec epochs using the SOMNOmedics PSG analysis software (Domino panel ver. 3.0.0.8) and manual editing. The setup for the polysomnography (PSG) involved the use of the Home-Sleep-Test REM+ device, which records various sleep parameters, including EEG, EOG, and EMG. EEG measurements will be obtained using silver/silver chloride electrode sets, placed in four specific locations that allow for the monitoring of key brain regions associated with sleep cycles. These locations will be selected based on the standardized 10/20 system to ensure accurate representation of the frontal, central, and occipital regions, facilitating a comprehensive analysis of the sleep architecture. The use of these electrodes provides high-fidelity recordings essential for evaluating both the depth and quality of sleep stages.

For EEG, the electrode will be positioned in the frontopolar region, specifically at Fp1 (left side) and M1, allowing for the monitoring of brain activity. The EOG electrodes will be placed near the left and right eyes to record eye movements, which is crucial for analyzing sleep stages, including REM sleep. The system is designed for ease of use: a tablet guides the patient through the sensor application process. Once the test begins, the tablet records data that the sensors transfer via Bluetooth. After the sleep study is completed, all data is automatically transferred from the tablet to a cloud platform for comprehensive analysis, ensuring seamless and accurate evaluation of sleep parameters such as brain activity, eye movements, and muscle tone. EEG analysis will be reported as follows: Total Sleep Time (total amount of sleep time scored during the total recording time); Sleep Efficiency (Total sleep time/Time in bed); Sustained Sleep Efficiency (Total sleep time/Time in bed - Sleep latency stage 2); Sleep Latency (the period of time it takes for a person to fall asleep after they have gone to bed and tried to initiate sleep); Sleep Latency N1 (the period of time between wakefulness and when sleep begins); Sleep Latency N2 (the period of time between time in bed and sleep onset stage 2); REM Latency (the amount of time elapsed between the onset of sleep to the first REM stage).

Handgrip strength assessment The handgrip test will be used for the assessment of maximum isometric strength of the hand and arm muscles (Marsden MG-4800 Hand Dynamometer) and used as a measurement of muscle tone alertness. Reduction of muscle strength after the intervention, was assessed as reduction of muscle tone.

Massage Sessions

Activation (Sports) massage The activation (sports) type of massage will be used as one of the massage interventions. This technique will be performed on a full body with more attention given to specific leg muscle groups such as the feet, the gastrocnemius, the femoral biceps and quadriceps and in upper body muscle groups such as the triceps, the rhomboid, the deltoid, the trapezius and head areas. Briefly, this type of massage involves a wide range of techniques that include effleurage, palmar sliding, pounding and hacking. The total duration of the activation message will be 30 minutes.

Relaxation massage The Relaxation type of massage will be used as the second type of intervention in this study. This technique is designed to promote deep relaxation, reduce stress and enhance overall well-being. It is characterized by the use of four primary techniques performed on the full body, including the palms and feet. Specifically, these techniques consist of effleurage (long, smooth, gliding strokes), petrissage (light pressure, rhythmic movements) and vibration gentle shaking movements. In addition to these, the technique also incorporates rhythmic movements and deep light pressure to enhance relaxation and alleviate tension. The total duration of the Relaxation massage will be 30 minutes.

Statistical Analysis The statistical analysis will be performed using IBM SPSS Statistics version 29 (SPSS Inc., Chicago, U.S.A.) An independent samples T-test will be used to examine differences in baseline characteristics and questionnaires between male and female subjects. A General Linear Model (GLM) Repeated Measures ANOVA will be used to assess changes in all parameters among the 3 different scenarios. A Bonferroni post-hoc test will be performed to assess individual differences. To assess normality, the Shapiro-Wilk test will be used alongside graphical representations, including the Normal Q-Q plot, Detrended Normal Q-Q plot, and Box Plot. The significance level is set at 5%. Beyond significance testing (p-value), effect size will also be considered to evaluate the magnitude of the effect.

Power Analysis Sample size calculations has been conducted using G*Power 3.1. The post-hoc "GLM" - Repeated measures, within factors" method was used to calculate the power analysis. The resulting minimum required sample size to achieve 85% power was 14 for 2-sided group-1 and group-2 errors 5% [(Effect size 0.60, Critical F 4.10, Ndf 2, Ddf 10, Power (1-β err pob) = 0.86 (86% power)].

ELIGIBILITY:
Inclusion Criteria:

• Complains of poor sleep assessed by Pittsburgh Quality Sleep Index score >5

Exclusion Criteria:

* history of mental illness,
* dermatological diseases,
* allergies to massage oil,
* history of epilepsy,
* acute or chronic condition that would limit the ability of the patient to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender at birth
Enrollment: 15 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Sleep Latency N1 | Sleep latency N1 will be calculated after the intervention (35 minutes after the initiation of the protocol)
  Sleep Latency N1 is the period of time between wakefulness and when sleep begins (stage 1)

SECONDARY OUTCOMES:
Relaxation Score | Relaxation score is assessed at baseline and after the intervention (35 minutes after the initiation of the protocol))
  The Relaxation score will be calculated by the Relaxation State Questionnaire assessing the state of relaxation before and after the intervention.
  The RSQ score ranges from 10 to 50 with a higher score implying a better outcome (the larger the number, the more relaxed is the person).

OTHER OUTCOMES:
Muscle Tone | Muscle tone will be assessed at baseline and after the intervention (35 minutes after the initiation of the protocol)
  Reduction in muscle strenght after the intervention is considered as reduction in muscle tone.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos Sakkas, PhD, Principal Investigator — University of Thessaly
Locations (1):
- School of Physical Education, Sports and Dietetics, TEFAA, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
Anonymized polysomnographic data will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2025 - June 2030
Access Criteria: Who: Academics or Researchers after a written request What: Raw data in SPSS format How: receive a link to download the data.
URL: https://www.dropbox.com/scl/fo/u1pi4s2nixxglh45qs5cp/AApyC4wkfSxleyXl9ido6O0?rlkey=7tvy059m6fy92w6hgmo1fk385&dl=0

REFERENCES:
- [Background] Dakic M, Toskic L, Ilic V, Duric S, Dopsaj M, Simenko J. The Effects of Massage Therapy on Sport and Exercise Performance: A Systematic Review. Sports (Basel). 2023 May 29;11(6):110. doi: 10.3390/sports11060110. PMID 37368560
- [Background] Guo J, Li L, Gong Y, Zhu R, Xu J, Zou J, Chen X. Massage Alleviates Delayed Onset Muscle Soreness after Strenuous Exercise: A Systematic Review and Meta-Analysis. Front Physiol. 2017 Sep 27;8:747. doi: 10.3389/fphys.2017.00747. eCollection 2017. PMID 29021762
- [Background] Simpson NS, Gibbs EL, Matheson GO. Optimizing sleep to maximize performance: implications and recommendations for elite athletes. Scand J Med Sci Sports. 2017 Mar;27(3):266-274. doi: 10.1111/sms.12703. Epub 2016 Jul 1. PMID 27367265
- [Background] Dutheil F, Danini B, Bagheri R, Fantini ML, Pereira B, Moustafa F, Trousselard M, Navel V. Effects of a Short Daytime Nap on the Cognitive Performance: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Sep 28;18(19):10212. doi: 10.3390/ijerph181910212. PMID 34639511
- [Derived] Ntoumas I, Karatzaferi C, Boubougiatzi F, Manakou N, Aslanidi A, Giannaki CD, Papanikolaou F, Dardiotis E, Lavdas E, Sakkas GK. Massage positively influences daytime brain activity and reduces arousal state in poor sleepers: a randomized controlled trial. BMC Complement Med Ther. 2025 Jul 28;25(1):290. doi: 10.1186/s12906-025-05022-6. PMID 40722019